CLINICAL TRIAL: NCT00873431
Title: An Open-Label Phase 1 Study Assessing the Safety, Immunogenicity and Dose Response of IC47, a New Vaccine Against Streptococcus Pneumoniae, in Healthy Subjects.
Brief Title: Open-Label Study Assessing The Safety, Immunogenicity and Dose Response of IC47
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IC47-101
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Pneumococcal Infections
Keywords: Prevention of pneumococcal infections
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IC47 30 mcg (Experimental): 30 mcg with Alum
  Interventions: Biological: IC47
- IC47 30 mcg w/o (Experimental): 30 mcg without Alum
  Interventions: Biological: IC47
- IC47 150 mcg (Experimental): 150 mcg with Alum
  Interventions: Biological: IC47
- IC47 150 mcg w/o (Experimental): 150 mcg without Alum
  Interventions: Biological: IC47

INTERVENTIONS:
Biological: IC47 — solution/suspension for i.m. injection dosage: 30/150 mcg frequency: 3 times at Day 0, Day 42 and Day 84

SUMMARY:
The main aim of this clinical study is to investigate the safety and tolerability of different dose strengths of IC47 up to 6 months after the first vaccination.

A total of 32 healthy subjects (male or female) will participate in this clinical study. The subjects will be divided into 4 groups of 8 subjects each. Thirty (30) μg or 150 μg of IC47 will be administered three times in intervals of 42 days each.

DETAILED DESCRIPTION:
This Phase 1 study will be conducted in four groups of 8 healthy subjects at a single study center. 32 subjects will be enrolled. The following table shows the design of the different study groups. The amount of protein shown in the table refers to the total protein content and is comprised of an equal amount of the three individual components.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Healthy adults ≥ 18 to </= 65
* female subjects: post-menopausal or practicing reliable methods of contraception during the study

Exclusion Criteria:

* History of autoimmune diseases and malignancies.
* History of severe hypersensitivity reactions and anaphylaxis.
* Immunodeficiency due to immunosuppressive therapy.
* Infection with HIV, Hepatitis B or Hepatitis C.
* Pregnancy, lactation
* Vulnerable subjects

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-03; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of any SAEs (possibly)related to the study vaccine | Day 0 - Day 264
Occurrence of any Grade 3 or higher adverse reactions (possibly)related to the study vaccine | Day 0 - Day 264
Occurrence of solicited local and systemic AEs within 1 week after vaccination | Day 0 - Day 264

SECONDARY OUTCOMES:
Determination of vaccine-specific IgG levels | Day 0 - Day 264

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Hatzenbichler, PhD, Study Director — Valneva Austria GmbH
Locations (1):
- Parexel International GmbH, Institute for Clinical Pharmacology, Berlin, State of Berlin, Germany